CLINICAL TRIAL: NCT02428309
Title: A Phase I, Open-Label, Dose Escalation Trial Exploring the Safety and Tolerability of Autologous Polyclonal Regulatory T Cell Therapy in Adults With Active Cutaneous Lupus (ALE08)
Brief Title: Autologous Polyclonal Tregs for Lupus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to participant recruitment feasibility
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ALE08
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic
Keywords: active cutaneous lupus; systemic lupus erythematosus (SLE); autologous polyclonal regulatory T cell Therapy; polyclonal Tregs for treatment of lupus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low Dose Treg Cohort (Experimental): 3-6 participants will receive a single infusion of 1 x 10^ 8 autologous polyclonal Tregs (ex vivo selected and expanded)
  Interventions: Biological: Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells
- Medium Dose Treg Cohort (Experimental): Sequential dose escalation, 3-6 subjects will receive a single infusion of 4 x 10^ 8 autologous polyclonal Tregs (ex vivo selected and expanded)
  Interventions: Biological: Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells
- High Dose Treg Cohort (Experimental): Sequential dose escalation, 3-6 participants will receive a single infusion of 16 x 10^ 8 autologous polyclonal Tregs (ex vivo selected and expanded)
  Interventions: Biological: Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells

INTERVENTIONS:
Biological: Ex vivo Expanded Human Autologous Polyclonal Regulatory T Cells
  Other Names: Ex vivo Expanded Autologous CD4+CD127lo/-CD25+ Polyclonal Regulatory T Cells

SUMMARY:
The primary purpose of this Phase 1 study is to evaluate the safety, tolerability, and effect of 3 different doses of Treg therapy in adults with skin (cutaneous) involvement of their lupus. Targeting cutaneous disease offers the ability to control background therapy, readily detect clinical effects, and perform research analyses not only in blood but also skin. Safety, disease activity, and mechanism of Tregs will be evaluated. The intent is to support dose selection for a future larger efficacy trial in lupus.

DETAILED DESCRIPTION:
The investigational therapy in this trial, regulatory T cells (Tregs), is evaluating an alternative to traditional immunosuppressive therapies for the treatment of systemic lupus erythematosus (SLE, lupus). Too frequently, aggressive therapies are inadequate in the control of the disease and have potent side effects and complications. The collection and expansion of one's own T cells harnesses a naturally occurring regulatory mechanism to restore self-tolerance in people with lupus. Tregs are a specialized subset of T cells that function to control the immune response. Studies have shown that in active lupus, the numbers and function of Treg cells are significantly decreased, which contributes to an overactive immune system and an increase in disease activity. The hope is that these naturally occurring Treg cells can be used for the treatment of autoimmune diseases, including lupus.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent.
* Diagnosis of SLE by American College of Rheumatology (ACR) criteria or biopsy proven primary cutaneous lupus.
* Presence of ≥ 2 active cutaneous lupus lesions based on (1) visual morphology and (2) at least a grade 2 erythema on CLASI activity score. Histopathologic confirmation is required unless the active lesions are of the same morphology to previously histologically proven cutaneous lupus lesions.
* The cutaneous lupus lesions must include any of the following subtypes:

  * Acute cutaneous lupus including maculopapular lupus rash and photosensitive lupus rash,
  * Subacute cutaneous lupus,
  * Chronic cutaneous lupus including discoid lupus and hypertrophic (verrucous) lupus,
  * Lupus timidus
* Positive test for Epstein-Barr virus (EBV) antibody.
* Adequate venous access to support draw of 400 mL whole blood and infusion of investigational therapy.

Exclusion Criteria:

* New onset of cutaneous lupus which has not been treated with broad spectrum sunscreen (UVA and UVB) in combination with either antimalarials or another systemic medication for at least 3 months.
* Prednisone dose > 15mg/day within the 30 days prior to screening.
* Addition of a new medication, or change in the dose of any background medication, used to treat any aspect of SLE. Specifically:

  * addition or change in systemic glucocorticoids, antimalarials, methotrexate, mycophenolate mofetil, mycophenolic acid, azathioprine, cyclosporine, tacrolimus, thalidomide, lenalidomide, dapsone, acitretin, or isotretinoin within 90 days prior to screening
  * treatment with cyclophosphamide within 90 days prior to screening.
* Doses of background medications at Screening visit:

  * hydroxychloroquine > 400 mg/day,
  * chloroquine > 250 mg/day,
  * quinacrine >100 mg/day,
  * methotrexate > 25 mg/week,
  * mycophenolate mofetil (MMF)> 3000 mg/day,
  * mycophenolic acid > 720 mg/day BID,
  * azathioprine > 200 mg/day,
  * cyclosporine > 5 mg/day divided BID,
  * tacrolimus > 6 mg/day
  * thalidomide > 300 mg/day,
  * lenalidomide > 10 mg/day,
  * dapsone > 250 mg/day,
  * acitretin > 50 mg/d (or > 1 mg/kg/day),
  * isotretinoin > 120 mg/d (or > 2 mg/kg/day).
* Intravenous immunoglobulin (IVIG), plasmapheresis, or leukopheresis within the 90 days prior to screening.
* Use of rituximab within the 12 months prior to screening.
* Change in dosing frequency, concentration, or applied surface area of topical steroids, tacrolimus, and/or pimecrolimus within 4 weeks prior to screening.
* Active severe central nervous system lupus.
* SELENA-SLEDAI's seizure, psychosis, organic brain syndrome, visual disturbance,cranial nerve disorder, lupus headache, cerebrovascular accident (CVA), vasculitis,arthritis, myositis, mucosal ulcers, pleurisy, pericarditis, and fever scores > 8 total.
* Active lupus nephritis (spot protein / creatinine ratio > 1.0 mg/mg).
* End stage renal disease (estimated glomerular filtration rate [eGFR] < 20 ml/min/1.73m^2 using the CKD-EPI equation [53]).
* Drug induced lupus.
* Hemoglobin < 10 g/dL.
* White blood cell (WBC) count < 2,500/ mm^3 (equivalent to < 2.5 x10^9/L).
* Lymphocyte count < 625/mm^3 (equivalent to < 0.625 x10^9/L).
* Absolute neutrophil count < 1,500/mm3 (equivalent to < 1.5 x10^9/L).
* Platelets < 75,000/mm^3 (equivalent to < 75 x 10^9/L).
* Liver function test (aspartate aminotransferase [AST], alanine aminotransferase [ALT], or alkaline phosphatase [ALK]) results that are ≥ 2 times the upper limit of normal (ULN).
* Direct bilirubin > ULN.
* Active bacterial, viral, fungal, or opportunistic infections requiring systemic antiinfective therapy.
* Presence of positive purified protein derivative tuberculin skin test (PPD, > 5mm induration [regardless of Bacille Calmette Guerin (BCG) vaccine administration]) or positive or indeterminate QuantiFERON(R)-TB Gold In-Tube Test (QFT-G_IT) at screening.
* Evidence of infection with human immunodeficiency virus (HIV), hepatitis B (as assessed by HBsAg and anti-HBc) or hepatitis C.
* Detectable circulating EBV or cytomegalovirus (CMV) genomes or active infection.
* Chronic infection that is currently being treated with suppressive anti-infective therapy, including but not limited to tuberculosis, pneumocystis, CMV, herpes zoster, and atypical mycobacteria.
* Herpes simplex virus infection requiring chronic, suppressive therapy with an anti-viral medication.
* Receipt of a live-attenuated vaccine within 12 months prior to screening.
* Concomitant malignancies or a history of malignancy, with the exception of adequately treated basal and squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
* Pregnancy.
* Breastfeeding.
* Unwilling or unable to use reliable method(s) of contraception from four weeks prior to Day 0 throughout three months after Treg dosing (males) or for two years after Treg dosing (females). Note: investigators of female participants of childbearing potential on concurrent MMF, and those participants themselves, whether or not they plan to become pregnant, are strongly encouraged to participate in Mycophenolate Risk Evaluation and Mitigation Strategy (REMS).
* Use of an experimental therapeutic agent within the calendar year prior to screening.
* Use of biologic medications other than rituximab within the 90 days or 5 half-lives,whichever is greater, prior to screening.
* Concomitant medical condition that places the subject at risk by participating in this study, including but not limited to:

  * another severe, systemic autoimmune disease or condition (besides lupus) requiring systemic immunosuppressive therapy (e.g., rheumatoid arthritis, systemic sclerosis, primary Sjogren's syndrome, primary vasculitis, psoriasis, multiple sclerosis, ankylosing spondylitis, and inflammatory bowel disease), or
  * severe, progressive, or poorly controlled renal, hepatic, hematological, gastrointestinal, pulmonary, cardiac, or neurological disease, either related or unrelated to SLE, or
  * history of significant infection or recurrent infection that, in the investigator's opinion, places the subject at risk by participating in this study
  * any other concomitant medical condition that, in the investigator's opinion, places the subject at risk by participating in this study.
* Comorbidities requiring glucocorticoid therapy, including those which have required three or more courses of systemic glucocorticoids within the previous 12 months.
* Current or history within the past year of substance abuse.
* Inability to comply with study and follow-up procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-08-27 (Actual); Primary Completion 2016-09-02 (Actual); Study Completion 2018-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dall'Era, MD, Study Chair — University of California, San Francisco; Anna Haemel, MD, Study Chair — University of California, San Francisco; Jeffrey Bluestone, PhD, Study Chair — University of California, San Francisco; Michael Rosenblum, MD, PhD, Study Chair — University of California, San Francisco; David Wofsy, MD, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan is to share participant level data and additional relevant materials in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts. Currently: study in progress-no data sharing.
Time Frame: The aim is to share data available to the public within 24 months upon completion of the study.
Access Criteria: Will be available to the public.
URL: http://www.immport.org/immport-open/public/home/home

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: Autoimmunity Centers of Excellence — http://www.autoimmunitycenters.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment occurred at one site in the United States. The site was activated in August 2015.
Groups:
- Dose 1 (1x10^8): Participant received a single infusion of 1 x 10^8 autologous polyclonal Tregs (ex vivo selected and expanded)
Period: Overall Study
Arm/Group | Dose 1 (1x10^8)
Started | 1
Completed | 1 (The enrolled participant completed treatment and was followed through week 152, per protocol.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participant received a single infusion of 1 x 10^8 autologous polyclonal Tregs (ex vivo selected and expanded).
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (NA) — One participant was enrolled in the study.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Significant Adverse Events (AEs) Through Week 48
Description: A significant adverse event is any related National Cancer Institute's Common Terminology Criteria for Adverse Events, Version 4.0 Grade 3 or higher AE or any related serious adverse event. Related is defined as being possibly, probably, or definitely related to the ex vivo expanded autologous PolyTregs, as determined by the safety review committee.
Time Frame: From time of signed informed consent to Week 48
Population: One participant enrolled in the study that received a single infusion of 1 x 10^8 autologous polyclonal Tregs (ex vivo selected and expanded)
Measure: Number; unit: Events
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Events | 0

2. Secondary Outcome: Number of Significant Adverse Events (AEs) Through Week 152
Description: as for outcome 1
Time Frame: From time of signed informed consent to Week 152
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Events | 0

3. Secondary Outcome: Number of Grade 3 or Higher Adverse Events (AEs) Through Week 152
Description: Adverse events (AEs) Grade 3 or higher were graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events, Version 4.0.
Time Frame: From time of signed informed consent to Week 152
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Events | 1

4. Secondary Outcome: Number of Infection-Related Adverse Events (AEs) Through Week 152
Description: If the adverse event was believed to be caused by a viral, bacterial, or fungal organism, regardless of whether it was treated with antibiotics or not, then it was classified as infection-related.
Time Frame: From time of signed informed consent to Week 152
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Events | 0

5. Secondary Outcome: Number of Lupus Flares Through Week 152 by Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) and Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) Criteria
Description: An activity score increase of ≥4 CLASI points defines a flare. A mild/moderate flare includes at least one of the following SELENA-SLEDAI criteria: Increase in the SLEDAI Score of ≥3 points, new or worse discoid, photosensitive, profundus, cutaneous vasculitis, bullous lupus, nasopharyngeal ulcers, pleuritic, pericarditis, arthritis, fever attributable to SLE; increase in prednisone (<0.5 mg/kg/day); added NSAID or Plaquenil; increase in PhGA (<2.5 [on a 3.0 indexed VAS scale]). A severe flare includes at least one of the following SELENA-SLEDAI criteria: Increase of >12 in the SLEDAI Score; new or worse CNS-SLE, vasculitis, nephritis, myositis, platelet count <60,000/mm^3, hemolytic anemia with hemoglobin <7% or decrease in hemoglobin >3%; prednisone >0.5 mg/kg/day; new Cyclophosphamide, Azathioprine, Methotrexate, Mycophenolate Mofetil, or hospitalization attributable to SLE; increase in PhGA to >2.5.
Time Frame: From time of signed informed consent to Week 152
Population: as for outcome 1
Measure: Number; unit: Flares
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Flares
  No.of lupus flares (CLASI) | 0
  No. of lupus flares (SELENA-SLEDAI) | 1

6. Secondary Outcome: Number Infusion-Related Adverse Events (AEs) Within 24 Hours of Infusion
Description: Any infusion-related adverse events Grade 1 or higher within 24 hours of polyclonal Treg infusion. This study graded the severity of adverse events according to the National Cancer Institute's Common Terminology Criteria for Adverse Events, Version 4.0.
Time Frame: From time of infusion to 24 hours post infusion
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Events | 0

7. Secondary Outcome: Change From Baseline: Alkaline Phosphatase (ALK), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST)
Description: Change=Post Baseline value minus Baseline value. A positive difference reflects an increased laboratory parameter value over time; a negative difference reflects a decreased laboratory parameter value over time. Normal laboratory values are based on subject age, gender, and the specific laboratory methods that were used to determine the lab values.
Time Frame: Baseline (Visit 0) and Weeks 4, 12, 48, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
U/L
  Alkaline Phosphatase (ALK) at Week 4 | -9 (NA) — Not applicable as only one participant was analyzed.
  Alkaline Phosphatase (ALK) at Week 12 | 4 (NA) — Not applicable as only one participant was analyzed.
  Alkaline Phosphatase (ALK) at Week 48 | 4 (NA) — Not applicable as only one participant was analyzed.
  Alkaline Phosphatase (ALK) at Week 152 | -2 (NA) — Not applicable as only one participant was analyzed.
  Alanine Aminotransferase (ALT) at Week 4 | -1 (NA) — Not applicable as only one participant was analyzed.
  Alanine Aminotransferase (ALT) at Week 12 | -3 (NA) — Not applicable as only one participant was analyzed.
  Alanine Aminotransferase (ALT) at Week 48 | -1 (NA) — Not applicable as only one participant was analyzed.
  Alanine Aminotransferase (ALT) at Week 152 | -1 (NA) — Not applicable as only one participant was analyzed.
  Aspartate Aminotransferase (AST) at Week 4 | -5 (NA) — Not applicable as only one participant was analyzed.
  Aspartate Aminotransferase (AST) at Week 12 | -5 (NA) — Not applicable as only one participant was analyzed.
  Aspartate Aminotransferase (AST) at Week 48 | -4 (NA) — Not applicable as only one participant was analyzed.
  Aspartate Aminotransferase (AST) at Week 152 | -6 (NA) — Not applicable as only one participant was analyzed.

8. Secondary Outcome: Change From Baseline in g/dL: Albumin, Hemoglobin
Description: Change=Post Baseline value minus Baseline value. A positive difference reflects an increased laboratory parameter value over time; a negative difference reflects a decreased laboratory parameter value over time. Normal laboratory values depend on a subject age, gender, and the specific laboratory methods that were used to determine the lab values.
Time Frame: Baseline (Visit 0) and Weeks 4, 12, 48, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
g/dL
  Albumin at Week 4 | NA (NA) — Not collected/available.
  Albumin at Week 12 | 0.4 (NA) — Not applicable as only one participant was analyzed
  Albumin at Week 48 | 0.2 (NA) — Not applicable as only one participant was analyzed
  Albumin at Week 152 | 0.2 (NA) — Not applicable as only one participant was analyzed
  Hemoglobin at Week 4 | 1.6 (NA) — Not applicable as only one participant was analyzed
  Hemoglobin at Week 12 | 1.5 (NA) — Not applicable as only one participant was analyzed
  Hemoglobin at Week 48 | 1.3 (NA) — Not applicable as only one participant was analyzed
  Hemoglobin at Week 152 | 1.0 (NA) — Not applicable as only one participant was analyzed

9. Secondary Outcome: Change From Baseline in mg/dL: Total Bilirubin, Creatinine
Description: as for outcome 8
Time Frame: Baseline (Visit 0) and Weeks 4, 12, 48, and 152
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: mg/dL
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
mg/dL
  Total Bilirubin at Week 4 | 0.1 (NA) — Not applicable as only one participant was analyzed
  Total Bilirubin at Week 12 | -0.2 (NA) — Not applicable as only one participant was analyzed
  Total Bilirubin at Week 48 | 0.0 (NA) — Not applicable as only one participant was analyzed
  Total Bilirubin at Week 152 | -0.2 (NA) — Not applicable as only one participant was analyzed
  Creatinine at Week 4 | 0.1 (NA) — Not applicable as only one participant was analyzed
  Creatinine at Week 12 | 0.0 (NA) — Not applicable as only one participant was analyzed
  Creatinine at Week 48 | 0.1 (NA) — Not applicable as only one participant was analyzed
  Creatinine at Week 152 | 0.1 (NA) — Not applicable as only one participant was analyzed

10. Secondary Outcome: Change From Baseline in mmol/L: Potassium, Sodium, Chloride
Description: as for outcome 8
Time Frame: Baseline (Visit 0) and Weeks 4, 12, 48, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
mmol/L
  Total Potassium at Week 4 | -0.2 (NA) — Not applicable as only one participant was analyzed
  Total Potassium at Week 12 | -0.4 (NA) — Not applicable as only one participant was analyzed
  Total Potassium at Week 48 | -0.3 (NA) — Not applicable as only one participant was analyzed
  Total Potassium at Week 152 | -0.7 (NA) — Not applicable as only one participant was analyzed
  Sodium at Week 4 | 4 (NA) — Not applicable as only one participant was analyzed
  Sodium at Week 12 | 2 (NA) — Not applicable as only one participant was analyzed
  Sodium at Week 48 | 3 (NA) — Not applicable as only one participant was analyzed
  Sodium at Week 152 | 5 (NA) — Not applicable as only one participant was analyzed
  Chloride at Week 4 | -1 (NA) — Not applicable as only one participant was analyzed
  Chloride at Week 12 | -2 (NA) — Not applicable as only one participant was analyzed
  Chloride at Week 48 | -3 (NA) — Not applicable as only one participant was analyzed
  Chloride at Week 152 | -1 (NA) — Not applicable as only one participant was analyzed

11. Secondary Outcome: Change From Baseline in Cell Counts: White Blood Cells (WBC), Total Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, Platelets
Description: as for outcome 8
Time Frame: Baseline (Visit 0) and Weeks 4, 12, 48, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cell Count X 10^9/L
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Cell Count X 10^9/L
  White Blood Cells (WBC) at Week 4 | 0.8 (NA) — Not applicable as only one participant was analyzed
  White Blood Cells (WBC) at Week 12 | 1.3 (NA) — Not applicable as only one participant was analyzed
  White Blood Cells (WBC) at Week 48 | 1.2 (NA) — Not applicable as only one participant was analyzed
  White Blood Cells (WBC) at Week 152 | 1.1 (NA) — Not applicable as only one participant was analyzed
  Total Neutrophils at Week 4 | 0.6 (NA) — Not applicable as only one participant was analyzed
  Total Neutrophils at Week 12 | 0.9 (NA) — Not applicable as only one participant was analyzed
  Total Neutrophils at Week 48 | 0.9 (NA) — Not applicable as only one participant was analyzed
  Total Neutrophils at Week 152 | 0.8 (NA) — Not applicable as only one participant was analyzed
  Lymphocytes at Week 4 | 0.3 (NA) — Not applicable as only one participant was analyzed
  Lymphocytes at Week 12 | 0.6 (NA) — Not applicable as only one participant was analyzed
  Lymphocytes at Week 48 | 0.2 (NA) — Not applicable as only one participant was analyzed
  Lymphocytes at Week 152 | 0.4 (NA) — Not applicable as only one participant was analyzed
  Monocytes at Week 4 | 0.1 (NA) — Not applicable as only one participant was analyzed
  Monocytes at Week 12 | 0.1 (NA) — Not applicable as only one participant was analyzed
  Monocytes at Week 48 | 0.3 (NA) — Not applicable as only one participant was analyzed
  Monocytes at Week 152 | 0.2 (NA) — Not applicable as only one participant was analyzed
  Total Eosinophils at Week 4 | -0.2 (NA) — Not applicable as only one participant was analyzed
  Total Eosinophils at Week 12 | -0.2 (NA) — Not applicable as only one participant was analyzed
  Total Eosinophils at Week 48 | -0.2 (NA) — Not applicable as only one participant was analyzed
  Total Eosinophils at Week 152 | -0.2 (NA) — Not applicable as only one participant was analyzed
  Basophils at Week 4 | 0.0 (NA) — Not applicable as only one participant was analyzed
  Basophils at Week 12 | 0.0 (NA) — Not applicable as only one participant was analyzed
  Basophils at Week 48 | 0.0 (NA) — Not applicable as only one participant was analyzed
  Basophils at Week 152 | 0.0 (NA) — Not applicable as only one participant was analyzed
  Platelets at Week 4 | 66 (NA) — Not applicable as only one participant was analyzed
  Platelets at Week 12 | 62 (NA) — Not applicable as only one participant was analyzed
  Platelets at Week 48 | 16 (NA) — Not applicable as only one participant was analyzed
  Platelets at Week 152 | 44 (NA) — Not applicable as only one participant was analyzed

12. Secondary Outcome: Change From Baseline Red Blood Cell Count
Description: as for outcome 8
Time Frame: Baseline (Visit 0) and Weeks 4, 12, 48, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Cell Count x10^12/L
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
Cell Count x10^12/L
  Red Blood Cell Count at Week 4 | 0.6 (NA) — Not applicable as only one participant was analyzed
  Red Blood Cell Count at Week 12 | 0.7 (NA) — Not applicable as only one participant was analyzed
  Red Blood Cell Count at Week 48 | 0.6 (NA) — Not applicable as only one participant was analyzed
  Red Blood Cell Count at Week 152 | 0.9 (NA) — Not applicable as only one participant was analyzed

13. Secondary Outcome: Change From Baseline in mm/hr: Sedimentation Rate (ESR)
Description: as for outcome 8
Time Frame: Baseline (Visit 0) and Weeks 4, 12, 48, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
mm/hr
  Sedimentation Rate (ESR) at Week 4 | 0 (NA) — Not applicable as only one participant was analyzed
  Sedimentation Rate (ESR) at Week 12 | 4 (NA) — Not applicable as only one participant was analyzed
  Sedimentation Rate (ESR) at Week 48 | 20 (NA) — Not applicable as only one participant was analyzed
  Sedimentation Rate (ESR) at Week 152 | 2 (NA) — Not applicable as only one participant was analyzed

14. Secondary Outcome: Change From Baseline in Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score
Description: The Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) is a validated, physician-based assessment tool used to measure cutaneous lupus severity. Severity is calculated based on disease activity (erythema and scale) and damage (dyspigmentation and scarring) for the cumulative areas of involved skin. Severity categories based on the CLASI activity score are as follows: mild (0-9), moderate (10-20), and severe (21-70). A 4-point or 20% change in the CLASI activity score identifies a clinically meaningful change. A 4-point increase in the CLASI activity score indicates a flare.
Time Frame: Baseline (Visit 0) and Weeks 12, 24, 36, 48, 100, 126, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
units on a scale
  Week 12 | -2 (NA) — Not applicable as only one participant was analyzed
  Week 24 | -1 (NA) — Not applicable as only one participant was analyzed
  Week 36 | -1 (NA) — Not applicable as only one participant was analyzed
  Week 48 | -1 (NA) — Not applicable as only one participant was analyzed
  Week 100 | -15 (NA) — Not applicable as only one participant was analyzed
  Week 126 | -10 (NA) — Not applicable as only one participant was analyzed
  Week 152 | -12 (NA) — Not applicable as only one participant was analyzed

15. Secondary Outcome: Change From Baseline in SELENA-SLEDAI Total Score
Description: The Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus (SLE) Disease Activity Index (SELENA-SLEDAI) score is a weighted scale score ranging from 0 to 105 based on the presence or absence of 24 manifestations of SLE. The SELENA-SLEDAI assesses disease activity for 10 days prior to and including the day of assessment. Positive change in the SELENA-SLEDAI score indicates increased disease activity.
Time Frame: Baseline (Visit 0) and Weeks 12, 24, 36, 48, 100, 126, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
units on a scale
  Week 12 | 0 (NA) — Not applicable as only one participant was analyzed
  Week 24 | 0 (NA) — Not applicable as only one participant was analyzed
  Week 36 | -2 (NA) — Not applicable as only one participant was analyzed
  Week 48 | -2 (NA) — Not applicable as only one participant was analyzed
  Week 100 | -2 (NA) — Not applicable as only one participant was analyzed
  Week 126 | 0 (NA) — Not applicable as only one participant was analyzed
  Week 152 | 0 (NA) — Not applicable as only one participant was analyzed

16. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PGA)
Description: The global assessment (PGA) is a visual 3-inch analog scale from 0 to 3 in which the participant marks the scale according to perceived disease activity. A score of 0 corresponds to no lupus disease activity and a score of 3 corresponds to severe disease activity. A positive change from baseline indicates more disease activity.
Time Frame: Baseline (Visit 0) and Weeks 12, 24, 36, 48, 100, 126, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
inches
  Week 12 | -0.625 (NA) — Not applicable as only one participant was analyzed
  Week 24 | -0.875 (NA) — Not applicable as only one participant was analyzed
  Week 36 | -0.625 (NA) — Not applicable as only one participant was analyzed
  Week 48 | 1.000 (NA) — Not applicable as only one participant was analyzed
  Week 100 | -1.000 (NA) — Not applicable as only one participant was analyzed
  Week 126 | 0.500 (NA) — Not applicable as only one participant was analyzed
  Week 152 | 0.000 (NA) — Not applicable as only one participant was analyzed

17. Secondary Outcome: Change From Baseline in Physician's Global Assessment (PhGA)
Description: The physician's global assessment (PhGA) is a visual analog 3-inch scale in the SELENA-SLEDAI that is scored from 0 to 3 by the physician. A score of 0 corresponds to no lupus disease activity and a score of 3 corresponds to severe disease activity. A positive change from baseline indicates more disease activity.
Time Frame: Baseline (Visit 0) and Weeks 12, 24, 36, 48, 100, 126, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
inches
  Week 12 | -0.125 (NA) — Not applicable as only one participant was analyzed
  Week 24 | -0.125 (NA) — Not applicable as only one participant was analyzed
  Week 36 | -0.125 (NA) — Not applicable as only one participant was analyzed
  Week 48 | -0.125 (NA) — Not applicable as only one participant was analyzed
  Week 100 | -0.938 (NA) — Not applicable as only one participant was analyzed
  Week 126 | 0.875 (NA) — Not applicable as only one participant was analyzed
  Week 152 | 0.563 (NA) — Not applicable as only one participant was analyzed

18. Secondary Outcome: Change From Baseline in Anti-dsDNA Antibody Titers
Description: Double-stranded DNA is one of multiple diagnostic tests for SLE and high levels may be associated with disease activity. The positive range is based on the normal range from the local laboratory. A positive change from baseline value indicates the detection of autoantibodies to double-stranded DNA.
Time Frame: Baseline ( Visit 0) and Weeks 12, 24, 36, 48, 100, 126, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
IU/mL
  Week 12 | 7 (NA) — Not applicable as only one participant was analyzed
  Week 24 | 35 (NA) — Not applicable as only one participant was analyzed
  Week 36 | 136 (NA) — Not applicable as only one participant was analyzed
  Week 48 | 25 (NA) — Not applicable as only one participant was analyzed
  Week 100 | 138 (NA) — Not applicable as only one participant was analyzed
  Week 126 | 283 (NA) — Not applicable as only one participant was analyzed
  Week 152 | -37 (NA) — Not applicable as only one participant was analyzed

19. Secondary Outcome: Change From Baseline in Serum C3 Complement Levels
Description: C3 is a blood test that measures the activity of the complement component 3 (C3) protein. The normal C3 range is 71 to 159 mg/dL. Those with active systemic lupus erythematosus (SLE) may have a lower-than-normal level of C3. A decrease in C3 level over time may indicate SLE disease activity.
Time Frame: Baseline (Visit 0) and Weeks 12, 24, 36, 48, 100, 126, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
mg/dL
  Week 12 | -2 (NA) — Not applicable as only one participant was analyzed
  Week 24 | 11 (NA) — Not applicable as only one participant was analyzed
  Week 36 | 11 (NA) — Not applicable as only one participant was analyzed
  Week 48 | -4 (NA) — Not applicable as only one participant was analyzed
  Week 100 | 8 (NA) — Not applicable as only one participant was analyzed
  Week 126 | -6 (NA) — Not applicable as only one participant was analyzed
  Week 152 | 0 (NA) — Not applicable as only one participant was analyzed

20. Secondary Outcome: Change From Baseline in Serum C4 Complement Levels
Description: C4 is a blood test that measures the activity of the complement component 4 (C4) protein. The normal range is 13 to 30 mg/dL. Individuals with active systemic lupus erythematosus (SLE) may have a lower-than-normal level of C4. A decrease in C4 level over time may indicate disease activity.
Time Frame: Baseline (Visit 0) and Weeks 12, 24, 36, 48, 100, 126, and 152
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dose 1 (1x10^8)
Number analyzed (Participants) | 1
mg/dL
  Week 12 | -1 (NA) — Not applicable as only one participant was analyzed
  Week 24 | -1 (NA) — Not applicable as only one participant was analyzed
  Week 36 | -3 (NA) — Not applicable as only one participant was analyzed
  Week 48 | -5 (NA) — Not applicable as only one participant was analyzed
  Week 100 | 1 (NA) — Not applicable as only one participant was analyzed
  Week 126 | -1 (NA) — Not applicable as only one participant was analyzed
  Week 152 | 3 (NA) — Not applicable as only one participant was analyzed

ADVERSE EVENTS:
Time Frame: From time of signed informed consent to Week 48.
Arm/Group | Dose 1 (1x10^8)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (1x10^8) (N=1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose 1 (1x10^8) (N=1)
Pericarditis (Cardiac disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study terminated early due to recruitment feasibility issues. One participant was enrolled, received polyclonal Treg treatment and was followed through week 152, per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No